CLINICAL TRIAL: NCT02890641
Title: Genetic and Electrophysiologic Study in Focal Drug-resistant Epilepsies
Acronym: GENEPHY
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GDR_2015_15
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Refractory Focal Epilepsy; Focal Cortical Dysplasia; Hemimegalencephaly; Tuberous Sclerosis; Mild Malformation of Cortical Development With Oligodendroglial Hyperplasia in Epilepsy (MOGHE)
Keywords: Focal Cortical Dysplasia; Cortical Malformation; Hemimegalencephaly; Tuberous sclerosis; Mild malformation of cortical development with oligodendroglial hyperplasia in epilepsy (MOGHE); Hypothalamic hamartomas; Refractory Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Focal Cortical Dysplasia; Hemimegalencephaly; Tuberous Sclerosis; Hypothalamic hamartomas

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cortical tissue removed during neurosurgical intervention for epilepsy

GROUPS / COHORTS (1):
- Children undergoing epilepsy surgery at the Rothschild Foundation, Paris.: Sequencing of paired blood-brain DNA samples
  Interventions: Genetic: Sampling of blood, frozen resected tissues, and cerebrospinal fluid (CSF)

INTERVENTIONS:
Genetic: Sampling of blood, frozen resected tissues, and cerebrospinal fluid (CSF) — Sampling of blood, frozen resected tissue, and cerebrospinal fluid (CSF); sequencing of paired blood-brain DNA samples

SUMMARY:
Brain somatic mutations in genes belonging to the mTOR signaling pathway are a frequent cause of cortical malformations, including focal cortical dysplasia and hemimegalencephaly, while SLC35A2 mutations are identified in MOGHE.

This study aims to identify brain somatic mutations in paired blood-brain samples and perform functional validation in children with drug-resistant focal epilepsy

ELIGIBILITY:
Inclusion Criteria:

* Children with focal drug-resistant epilepsy including Focal Cortical Dysplasia, Hemimegalencephaly, Tuberous Sclerosis, Mild malformation of cortical development with oligodendroglial hyperplasia in epilepsy (MOGHE), Hypothalamic Hamartomas, Sturge-Weber syndrome, Rasmussen encephalitis, gliomas)
* Their parents who have signed informed consent 1) for their child's participation (for parents) and 2) for themselves
* Social security coverage or foreign regime recognized in France

Exclusion Criteria:

* refusal to participate in the study
* contraindication to anaesthesia, to MRI or to surgery
* no medical insurance coverage

Ages: 3 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with focal drug-resistant epilepsy undergoing epilepsy surgery and their parents
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2015-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
qualitative genetic analysis | baseline
  Detection of brain somatic mutations and functional studies

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde CHIPAUX, MD, Principal Investigator — Fondation A de Rothschild; Stephanie Baulac, PhD, Study Chair — Institut du Cerveau et de la Moelle Epinière
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschld, Paris, France

REFERENCES:
- [Result] Baldassari S, Ribierre T, Marsan E, Adle-Biassette H, Ferrand-Sorbets S, Bulteau C, Dorison N, Fohlen M, Polivka M, Weckhuysen S, Dorfmuller G, Chipaux M, Baulac S. Dissecting the genetic basis of focal cortical dysplasia: a large cohort study. Acta Neuropathol. 2019 Dec;138(6):885-900. doi: 10.1007/s00401-019-02061-5. Epub 2019 Aug 23. PMID 31444548
- [Result] Bonduelle T, Hartlieb T, Baldassari S, Sim NS, Kim SH, Kang HC, Kobow K, Coras R, Chipaux M, Dorfmuller G, Adle-Biassette H, Aronica E, Lee JH, Blumcke I, Baulac S. Frequent SLC35A2 brain mosaicism in mild malformation of cortical development with oligodendroglial hyperplasia in epilepsy (MOGHE). Acta Neuropathol Commun. 2021 Jan 6;9(1):3. doi: 10.1186/s40478-020-01085-3. PMID 33407896
- [Result] Lee WS, Baldassari S, Chipaux M, Adle-Biassette H, Stephenson SEM, Maixner W, Harvey AS, Lockhart PJ, Baulac S, Leventer RJ. Gradient of brain mosaic RHEB variants causes a continuum of cortical dysplasia. Ann Clin Transl Neurol. 2021 Feb;8(2):485-490. doi: 10.1002/acn3.51286. Epub 2021 Jan 12. PMID 33434304
- [Result] Kim S, Baldassari S, Sim NS, Chipaux M, Dorfmuller G, Kim DS, Chang WS, Taly V, Lee JH, Baulac S. Detection of Brain Somatic Mutations in Cerebrospinal Fluid from Refractory Epilepsy Patients. Ann Neurol. 2021 Jun;89(6):1248-1252. doi: 10.1002/ana.26080. Epub 2021 Apr 20. PMID 33834539
- [Result] Barba C, Blumcke I, Winawer MR, Hartlieb T, Kang HC, Grisotto L, Chipaux M, Bien CG, Hermanovska B, Porter BE, Lidov HGW, Cetica V, Woermann FG, Lopez-Rivera JA, Canoll PD, Mader I, D'Incerti L, Baldassari S, Yang E, Gaballa A, Vogel H, Straka B, Macconi L, Polster T, Grant GA, Krskova L, Shin HJ, Ko A, Crino PB, Krsek P, Lee JH, Lal D, Baulac S, Poduri A, Guerrini R; SLC35A2 Study Group. Clinical Features, Neuropathology, and Surgical Outcome in Patients With Refractory Epilepsy and Brain Somatic Variants in the SLC35A2 Gene. Neurology. 2023 Jan 31;100(5):e528-e542. doi: 10.1212/WNL.0000000000201471. Epub 2022 Oct 28. PMID 36307217
- [Result] Checri R, Chipaux M, Ferrand-Sorbets S, Raffo E, Bulteau C, Rosenberg SD, Doladilhe M, Dorfmuller G, Adle-Biassette H, Baldassari S, Baulac S. Detection of brain somatic mutations in focal cortical dysplasia during epilepsy presurgical workup. Brain Commun. 2023 Jun 1;5(3):fcad174. doi: 10.1093/braincomms/fcad174. eCollection 2023. PMID 37324239
- [Result] Ribierre T, Bacq A, Donneger F, Doladilhe M, Maletic M, Roussel D, Le Roux I, Chassoux F, Devaux B, Adle-Biassette H, Ferrand-Sorbets S, Dorfmuller G, Chipaux M, Baldassari S, Poncer JC, Baulac S. Targeting pathological cells with senolytic drugs reduces seizures in neurodevelopmental mTOR-related epilepsy. Nat Neurosci. 2024 Jun;27(6):1125-1136. doi: 10.1038/s41593-024-01634-2. Epub 2024 May 6. PMID 38710875
- [Result] Sanders MWCB, Koeleman BPC, Brilstra EH, Jansen FE, Baldassari S, Chipaux M, Sim NS, Ko A, Kang HC, Blumcke I, Lal D, Baulac S, Lee JH, Aronica E, Braun KPJ. Somatic variant analysis of resected brain tissue in epilepsy surgery patients. Epilepsia. 2024 Dec;65(12):e209-e215. doi: 10.1111/epi.18148. Epub 2024 Oct 26. PMID 39460693
- [Result] Baldassari S, Klingler E, Teijeiro LG, Doladilhe M, Raoux C, Roig-Puiggros S, Bizzotto S, Couturier J, Gilbert A, Sami L, Ribierre T, Aronica E, Adle-Biassette H, Chipaux M, Jabaudon D, Baulac S. Single-cell genotyping and transcriptomic profiling of mosaic focal cortical dysplasia. Nat Neurosci. 2025 May;28(5):964-972. doi: 10.1038/s41593-025-01936-z. Epub 2025 Apr 30. PMID 40307383
- See also: Related Info — https://www.nlm.nih.gov/